CLINICAL TRIAL: NCT03246815
Title: STD Testing in Outpatient Practices-The STOP STDs Study
Brief Title: STD Testing in Outpatient Practices
Acronym: STOP
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: CDC Foundation (Other)
Responsible Party: Principal Investigator, Harold Wiesenfeld, Principal Investigator, University of Pittsburgh
Other Study IDs: PRO14110416
Record Dates: First submitted 2017-07-18; First posted 2017-08-11 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: STD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- universal opt-out screening for STDs: Patients who present to primary care practices who employee a universal opt-out strategy to medical assistants or nurses
- without universal opt-out screening for STDs: Patients who present to primary care practices who do not employee a universal opt-out strategy to medical assistants or nurses

SUMMARY:
National guidelines have recommended routine STD screening (chlamydia and gonorrhea) for sexually active young women under the age of 25. Despite these recommendations, many young women are not being screened for STDs, with some estimates that less than 50% of women receiving health care are screened for chlamydia. Untreated STDs can lead to important sequelae to women's reproductive health including pelvic inflammatory disease, infertility and ectopic pregnancy. One of the most important barriers to widespread STD screening is provider failure to recognize an opportunity for STD screening. The goal of this study is to determine whether offering STD screening (chlamydia and gonorrhea) by a non-physician member of the medical practice (who receives an automated alert indicating STD screening should be offered) will be associated with a higher rate of STD screening in young women attending primary care practices compared to usual care (where a physician offers screening with no electronic alert). This study will be performed in UPMC-affiliated primary care practices (Family Practice, Internal Medicine, OB/GYN, Pediatrics). Practices will be assigned to the intervention or usual care. The intervention will be an auto-task in the electronic medical record to the non-physician/NP/PA medical staff (medical assistants, LPNs, RNs) to offer chlamydia and gonorrhea screening via urine or self-collected vaginal sampling, in an opt-out manner, to eligible women. Practices assigned to the usual care group will not have the intervention. STD screening rates (# women undergoing STD screening/# eligible women) will be compared between the to groups (intervention practices and control practices). Results of this study may be important to guide national STD screening recommendations and will address critical barriers to widespread STD screening.

ELIGIBILITY:
Inclusion Criteria:

Women ages 15-24 Sexually Active Receiving care in one of the primary care offices affiliated with UPMC selected for this study.

Exclusion Criteria:

Pregnancy

Ages: 15 Years to 24 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Young women at risk for STDs
Sampling Method: Non-Probability Sample
Enrollment: 6771 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of STD Screening | Day 1
  Rate of screening (Chlamydia and Gonorrhea) in young women attending primary care practices
Number of Chlamydia and Gonorrhea infections identified | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Harold C Wiesenfeld, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC/associated community clinics, Pittsburgh, Pennsylvania, United States